CLINICAL TRIAL: NCT00001319
Title: Evaluation of the Epidemiology, Clinical Manifestations, Etiologies, and Immunology of Human Immunodeficiency Virus (HIV) Negative CD4 T Lymphocyte Deficient Patients
Brief Title: Evaluation of HIV-Negative Patients With Low CD4+ T Lymphocyte Counts
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920256; 92-I-0256
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-07

CONDITIONS: CD4 Lymphocytopenia; Idiopathic CD4 Positive T Lymphocytopenia
Keywords: HIV Negative; CD4 Deficiency; Retrovirus
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive

SUMMARY:
This study will evaluate HIV-negative patients with unusually low levels of CD4+ T lymphocytes (a type of white blood cell) to learn more about the clinical symptoms, cause, immunology, and biology of this problem. CD4+ T lymphocytes play an important role in immune function, and low counts may leave people susceptible to unusual infections. CD4+ T cell deficiencies are most often associated with HIV infection.

Patients 8 years of age and older with CD4+ T cell counts below 300 cells/mm3 who test negative for HIV infection by standard blood tests may be eligible for this study. Patients' family members and partners may also be enrolled to investigate the possible role of a genetic factor or exposure to some agent in this problem.

Patients will be evaluated at the NIH Clinical Center at least once, and generally two or more times. The evaluations, which may be done on an inpatient or outpatient basis, will include some or all of the following tests and procedures:

* Complete physical examination.
* Medical history, including questions about sexual contacts, intravenous drug use, travel, blood transfusions, previous illnesses, including sexually transmitted diseases, and health of family members.
* Urine test.
* Blood tests for routine and research purposes, including tests for HIV, hepatitis, syphilis and other infections, evaluation of immune function, and culture for viruses in the HIV family. No more than 1 pint of blood will be drawn every 6 weeks.
* Pregnancy test for women of childbearing potential.
* Skin tests for tuberculosis and immune function. These tests involve injecting a small amount of the substance to be tested just under the skin and looking for a raised area 1 to 2 days later.
* Apheresis. Whole blood is collected through an arm vein (similar to donating blood), and circulated through a cell separator machine, where it is spun to separate the components. The red cells are then returned to the patient either through the same needle or through a needle in the other arm, and the plasma and white cells are extracted for study. The procedure, which takes 1 to 2 hours, may be repeated up to 3 times.

Family members will have 60 cc (4 tablespoons) of blood drawn to determine CD4+ T cell counts.

DETAILED DESCRIPTION:
Low CD4+ T-cells in the absence of known etiology has been called idiopathic CD4+ T lymphocytopenia, and a case definition was established by the CDC as a CD4 count less than 300 cells/mL on 2 consecutive samples in a patient uninfected by HIV and with no other disease or treatment that might provide a reasonable alternative explanation for CD4 lymphocytopenia. Early investigations centered on a search for a novel retrovirus, but we and others have not found evidence of such a retrovirus. The patients that we have seen are heterogeneous, and it appears likely that there will be multiple etiologies for this syndrome. We are currently continuing to follow subjects long term and to see new subjects in order to continue to characterize the clinical aspects of patients who meet the case definition; to determine the natural history of ICL, and to provide samples to researchers who are interested in investigations into the pathogenesis of ICL.

ELIGIBILITY:
INCLUSION CRITERIA

Adults greater than or equal to 18 years of age.

CD4 count less than 300 cells/mmL on 2 consecutive samples.

Uninfected by HIV as determined by ELISA with confirmatory Western Blot

Absence of disease or treatment that might provide a reasonable alternative explanation for the CD4 cell count or might confound the evaluation. Examples of such diseases would be any acute, severe medical illness that had not resolved when CD4 cell counts were obtained; active tuberculosis; leukemia or lymphoma; or previously characterized immunodeficiency disorder. Treatment that that might provide a reasonable alternative explanation includes chemotherapy over a field that could affect bone marrow or supraphysiologic glucocorticoid therapy.

Capable of providing informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1992-09; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Roger PM, Bernard-Pomier G, Counillon E, Breittmayer JP, Bernard A, Dellamonica P. Overexpression of Fas/CD95 and Fas-induced apoptosis in a patient with idiopathic CD4+ T lymphocytopenia. Clin Infect Dis. 1999 May;28(5):1012-6. doi: 10.1086/514739. PMID 10452627
- [Background] Cunningham-Rundles C, Murray HW, Smith JP. Treatment of idiopathic CD4 T lymphocytopenia with IL-2. Clin Exp Immunol. 1999 May;116(2):322-5. doi: 10.1046/j.1365-2249.1999.00886.x. PMID 10337025
- [Background] Aldrich J, Gross R, Adler M, King K, MacGregor RR, Gluckman SJ. The effect of acute severe illness on CD4+ lymphocyte counts in nonimmunocompromised patients. Arch Intern Med. 2000 Mar 13;160(5):715-6. doi: 10.1001/archinte.160.5.715. No abstract available. PMID 10724063
- [Derived] Zonios DI, Falloon J, Bennett JE, Shaw PA, Chaitt D, Baseler MW, Adelsberger JW, Metcalf JA, Polis MA, Kovacs SB, Kovacs JA, Davey RT, Lane HC, Masur H, Sereti I. Idiopathic CD4+ lymphocytopenia: natural history and prognostic factors. Blood. 2008 Jul 15;112(2):287-94. doi: 10.1182/blood-2007-12-127878. Epub 2008 May 2. PMID 18456875